CLINICAL TRIAL: NCT04498559
Title: Evaluating Patient Knowledge of Pain Management and Safe Opioid Use Before Surgery
Brief Title: Patient Knowledge on Pain Management and Safe Opioid Use
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-2246
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Opioid Use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing total hip replacement: Patients at HSS Main Campus undergoing primary total hip replacement surgery, age range between 18 and 80 years old, and English speaking

SUMMARY:
The purpose of this study is to examine what patients currently know about opioids, including their role in pain management, side effects, risks of abuse, and proper storage and disposal. It is critical for patients to be properly informed about opioid usage in treating postoperative pain, but current gaps in patient knowledge are not well understood.

This study will help identify knowledge deficiencies and guide future patient education. Additionally, this study will examine possible patient factors that may be associated with these gaps. Evaluation of patient knowledge will be assessed through interviews conducted before patients' day of surgery.

DETAILED DESCRIPTION:
Opioids are frequently prescribed to treat pain after surgery, and while these medications may be effective analgesics they are also susceptible to misuse and addiction. There are growing concerns that prescription opioids contribute to the existing opioid supply and become potential sources for abuse1,2. In fact, opioids are often abused by those using medications not prescribed to them but obtained from friends or relatives3,4.

Many patients who undergo surgery are not given adequate information about opioids and strategies for postoperative pain management. Studies find that inadequate knowledge and inability to recall postoperative pain regimens result in poor compliance5. Many patients are also unaware of how to properly store and dispose of prescription opioids1,6 and this predisposes them to opioid misuse and improper saving and sharing of pills6.

Little is known, however, about the specific gaps in knowledge and what patient demographics may be associated with lack of understanding. As an initial step toward addressing these issues, this study seeks to identify deficiencies in patient understanding of opioids and pain management.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 80 years old
* Undergoing primary total hip replacement surgery
* English speaking

Exclusion Criteria:

* Medical background (profession that involves the prescribing, dispensing, handling, or administering of opioids)
* History of chronic opioid use (continuous opioid use for 3 or more months)
* Opioid use within the past 3 months
* Non-English speakers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total hip replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Patient's knowledge about opioids based on a qualitative assessment | Prior to surgery
  Patient's answers to opioid-related questions will be summarized using grounded theory, and a comparative analytic strategy to categories. A PI-provided scoring manual will also be used to quantify the accuracy and level of patients' knowledge about opioids. Reference: Berkwits M, Inui TS. Making use of qualitative research techniques. J Gen Intern Med. 1998;13(3):195-199. doi:10.1046/j.1525-1497.1998.00054.x

SECONDARY OUTCOMES:
Age | Prior to surgery
  Is the age the of patient associated with patients' knowledge of opioids
Sex | Prior to surgery
  Is the sex of the patient associated with patients' knowledge of opioids
Race | Prior to surgery
  Is the race of the patient associated with patients' knowledge of opioids
Ethnicity | Prior to surgery
  Is the ethnicity of the patient associated with patients' knowledge of opioids
Previous surgeries | Prior to surgery
  Are previous surgeries of the patient associated with patients' knowledge of opioids
Previous opioid usage | Prior to surgery
  Is the previous opioid usage of patient associated with patients' knowledge of opioids
Education level | Prior to surgery
  Is the education level of the patient associated with patients' knowledge of opioids
Occupation | Prior to surgery
  Is the occupation of the patient associated with patients' knowledge of opioids
Alcohol and tobacco use | Prior to surgery
  Is the alcohol and tobacco use of the patient associated with patients' knowledge of opioids

CONTACTS AND LOCATIONS:
Overall Officials: Bradley H Lee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 36 months after publication
Access Criteria: Researchers who provide methodologically sound proposal
  To achieve aims in the approved protocol
  Proposals should be directed to leeb@hss.edu. Proposals may be submitted up to 36 months after article publication. To gain access, data requestors will need to sign a data access agreement.